CLINICAL TRIAL: NCT00717951
Title: A Randomised,Multi-Center Study of Docetaxol Plus Capecitabine or Cisplatin in Anthracycline-Pretreated Patients With Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Academy Military Medical Science, China (Industry)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Zefei Jiang, Binghe,Xu, Academy Millitary Medical Science, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAX625; CBCSG003
Record Dates: First submitted 2008-07-14; First posted 2008-07-18 (Estimated); Last update posted 2008-07-25 (Estimated); Status verified 2008-05

CONDITIONS: Advanced Breast Cancer
Keywords: advanced breast cancer; docetaxol; capecitabine; cisplatin
MeSH Terms: interventions — Docetaxel; Cisplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Arm A is "docetaxol+capecitabine" chemotherapy
  Interventions: Drug: docetaxol, cisplatin, capecitabine
- B (Experimental): Arm B is "docetaxol+cisplatin" chemotherapy
  Interventions: Drug: docetaxol, cisplatin, capecitabine

INTERVENTIONS:
Drug: docetaxol, cisplatin, capecitabine — docetaxol(75mg/m2 d1 every 21 days) combined with cisplatin(75mg/m2 d1 every 21 days) VS docetaxol( 75mg/m2 d1 every 21 days) combined with capecitabine(2000mg/m2 d1-14 every 21 days)

SUMMARY:
Docetaxol plus capecitabine regimen is the standard treatment for the anthracycline-pretreated patients with advanced breast cancer. Cisplatin is an important drug for advanced breast cancer and potential effective drug for triple negative breast cancer.The study primary objective:Assess ORR,TTP,TTF and 2 year PFS rate between docetaxol+capecitabine and docetaxol+cisplatin.

The second objective:Assess the safety and QOL.

DETAILED DESCRIPTION:
The study main inclusion criteria are:1.age≥18,KPS>70.2.anthracycline-pretreated patients with advanced breast cancer.3.at least 1 measurable lesion as defined by modified RECIST criteria.4.screening laboratory values within the following parameters:ANC ≥1.5×109/L,Hemoglobin≥10.0 g/dl，Platelet≥100×109/L. 5. signed ICF The patients will be randomised two group: docetaxol+capecitabine and docetaxol+cisplatin. According to AE, the dose will be adjusted.

ELIGIBILITY:
Inclusion Criteria:

* age≥18y
* KPS≥ 70
* pathologic diagnosis of breast cancer
* at least 1 measurable lesion as defined by modified RECIST criteria
* screening laboratory values with the following parameters: hemoglobin:≥10.0 g/dl absolute neutrophils count:≥1.5×109/L platelet:≥100×109/L creatinine clearance rate: ≥60ml/min total bilirubin: ≤1.5 ×upper limits of normal Alkaline phosphatase,Aspartate aminotransferase and Alanine aminotransferase:≤ 2.5×upper limits of normal（≤5×upper limits of normal if liver metastasis are present)
* signed ICF
* for women of child bearing potential,a negative serum or urine pregnancy test result before study entry.

Exclusion Criteria:

* More than 2 cytotoxic chemotherapy treatment regimens for metastatic disease.
* prior exposure to 5-Fluorouracil continuous infusion.
* prior exposure docetaxol for metastatic disease
* Any other cancer within 5 years prior to screening with the exception of contralateral breast cancer,adequately treated cervical carcinoma in situ,or adequately treated basal or squamous cell carcinoma of skin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
ORR,TTP,TTF and 2 year PFS | 2008-2010

SECONDARY OUTCOMES:
safety and QOL | 2008-2010

CONTACTS AND LOCATIONS:
Overall Officials: jiang zefei, Ph.D, Principal Investigator — Academy MMS,China

REFERENCES:
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241
- [Derived] Egger SJ, Chan MMK, Luo Q, Wilcken N. Platinum-containing regimens for triple-negative metastatic breast cancer. Cochrane Database Syst Rev. 2020 Oct 21;10(10):CD013750. doi: 10.1002/14651858.CD013750. PMID 33084020